CLINICAL TRIAL: NCT02357966
Title: A Phase I-II Study of the Safety and Efficacy of a True Human Antibody, 514G3, in Subjects Hospitalized With Bacteremia Due to Staphylococcus Aureus
Brief Title: Safety & Efficacy of True Human Antibody, 514G3, in Staphylococcus Aureus Bacteremia Hospitalized Subjects.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-PT029
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Staphylococcus Aureus, Bacteremia, Hospitalization, Antibody
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia

STUDY DESIGN:
Intervention Model Description: This is a Phase I/II, double blind placebo controlled trial of the True Human monoclonal antibody 514G3 in subjects hospitalized with Staphylococcus Aureus bacteremia.
  A phase I of the trial is a dose escalation study intended to assess the possible toxicity and to determine the recommended phase 2 dose of the study drug (514G3). Eligible subjects will be randomized (3:1) to receive single dose of 514G3 (Either 2, 10, 40 mg/kg) plus standard IV antibiotic therapy or single dose of placebo plus standard IV antibiotic therapy.
  A phase 2 of the trial is designed to assess the preliminary efficacy through randomization of subjects in two arm groups i.e. a single dose of 514G3 administered at the RP2D with standard IV treatment or placebo plus standard IV treatment.
  Eligible subjects will be randomized (2:1) to receive either a single dose of 514G3 plus standard IV antibiotic therapy versus a single dose of placebo plus standard IV antibiotic treatment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): A phase I of the trial is a dose escalation study intended to assess the possible toxicity and to determine the recommended phase 2 dose (RP2D) of the study drug (514G3).
  Randomized subjects were administered the study drug at 3 dose levels i.e. 2 mg/kg, 10 mg/kg, and 40 mg/kg or placebo.
  Interventions: Biological: 514G3 (2 mg/kg) plus standard IV antibiotic treatment; Biological: 514G3 (10 mg/kg) plus standard IV antibiotic treatment; Biological: 514G3 (40 mg/kg) plus standard IV antibiotic treatment; Other: Placebo plus standard IV antibiotic treatment
- Phase II (Experimental): A phase 2 of the trial is a dose expansion study designed to assess the preliminary efficacy. Eligible subjects are randomized (2:1) and received a single dose of 40 mg/kg study drug (514G3) with standard IV treatment versus placebo with standard IV treatment.
  Interventions: Biological: 514G3 (40 mg/kg) plus standard IV antibiotic treatment: Phase II; Other: Placebo plus standard IV antibiotic treatment: Phase II

INTERVENTIONS:
Biological: 514G3 (2 mg/kg) plus standard IV antibiotic treatment
  Other Names: True Human Monoclonal Antibody
  Arms: Phase I
Biological: 514G3 (10 mg/kg) plus standard IV antibiotic treatment
  Other Names: True Human Monoclonal Antibody
  Arms: Phase I
Biological: 514G3 (40 mg/kg) plus standard IV antibiotic treatment
  Other Names: True Human Monoclonal Antibody
  Arms: Phase I
Other: Placebo plus standard IV antibiotic treatment — Sterile isotonic formulation buffered at pH 6.2 - 6.5 plus standard IV antibiotic treatment
  Other Names: True Human Monoclonal Antibody
  Arms: Phase I
Biological: 514G3 (40 mg/kg) plus standard IV antibiotic treatment: Phase II — A single dose of 514G3 plus standard IV antibiotic therapy
  Other Names: True Human Monoclonal Antibody
  Arms: Phase II
Other: Placebo plus standard IV antibiotic treatment: Phase II — A single dose of placebo plus standard IV antibiotic therapy
  Other Names: True Human Monoclonal Antibody
  Arms: Phase II

SUMMARY:
This study is a Phase I/II, double-blind, placebo-controlled trial investigating the True Human monoclonal antibody 514G3 in subjects hospitalized with Staphylococcus aureus bacteremia. Phase I involves dose escalation to evaluate potential toxicity and establish the recommended phase 2 dosage of 514G3. In Phase II (dose expansion), eligible subjects will be randomized at a ratio of 2:1 to receive either a single dose of 514G3 with standard IV antibiotic therapy or a single dose of placebo with standard IV antibiotic therapy, aiming to assess safety and tolerability. The trial aims to determine the safety, efficacy, and optimal dosage regimen of 514G3 in these hospitalized subjects.

DETAILED DESCRIPTION:
The Phase I/II trial aims to assess the safety and efficacy of True Human monoclonal antibody 514G3 in hospitalized subjects with Staphylococcus aureus bacteremia.

Phase I entails dose escalation, with subjects randomized (3:1) at three dose levels of the study drug (2 mg/kg, 10 mg/kg, and 40 mg/kg) and placebo, utilizing central randomization. Dose-limiting toxicities (DLTs), defined as Grade 3 or greater adverse events related to 514G3 during follow-up, guide escalation. The Maximum Tolerated Dose (MTD) is determined based on DLT occurrence.

Phase II, focusing on preliminary efficacy, randomizes eligible subjects (2:1) to receive 514G3 or placebo with standard IV antibiotic therapy. Safety and efficacy assessments are conducted for both phases, encompassing pooled data from both the study drug and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. One or more blood cultures positive for staphylococcus aureus within 2 days of initiating treatment with 514G3.
2. Temperature ≥ 38.0°C
3. Age ≥18, male or female subjects.
4. Adequate renal function, defined by serum creatinine ≤ 2 times the upper limit of normal (ULN).
5. Adequate hepatic function
6. Adequate bone marrow function
7. For women of childbearing potential (WOCBP), a negative serum pregnancy test result at Screening.
8. Signed and dated institutional review board (IRB)/ Ethics Committee (EC)-approved informed consent before any protocol-specific screening procedures are performed.
9. Expected survival of at least 2 months.

Exclusion Criteria:

1. Polymicrobial bacteremia.
2. Known or suspected osteomyelitis or meningitis.
3. Patients that are being mechanically ventilated as a result of a pulmonary infection at the time of screening. Mechanical ventilation for other reasons, such as trauma, is acceptable.
4. Presence of any removable infection source (e.g., intravascular line, abscess, or prosthesis) that will not be removed or debrided within 3 days after randomization.
5. Definite or possible left-sided endocarditis, by Modified Duke Criteria, based on screening echocardiogram. Subjects with suspected right-sided endocarditis are permitted.
6. Need for emergent valve surgery at the time of screening, and/or the presence of decompensated heart failure or cardiogenic shock.
7. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
8. Infection with human immunodeficiency virus (HIV) and a CD4 count <200 cells/mm3.
9. Subjects with history of hypersensitivity to compounds of similar chemical or biologic composition to 514G3 or any component of its formulations.
10. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rupp, M.D., Study Chair — University of Nebraska
Locations (2):
- United States (2):
  - XBiotech Investigative Site, Columbus, Georgia
  - XBiotech Investigative Site, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data integrity and confidentiality

RESULTS

PARTICIPANT FLOW:
Groups:
- 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy: Participants received a single dose of 5143G (dose 2 mg/kg) plus standard IV antibiotic therapy.
- 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy: Participants received a single dose of 5143G (dose 10 mg/kg) plus standard IV antibiotic therapy.
- 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy: Participants received a single dose of 5143G (dose 40 mg/kg) plus standard IV antibiotic therapy.
- Placebo Plus Standard IV Antibiotic Therapy: Participants in this group received a single dose of placebo plus standard IV antibiotic therapy. Placebo is a sterile isotonic formulation buffered at pH 6.2 - 6.5
- Phase II: 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy: Participants received a single dose of 5143G (dose 40 mg/kg) plus standard IV antibiotic treatment
- Phase II: Placebo Plus Standard IV Antibiotic Therapy: Participants received a single dose of placebo plus standard IV antibiotic therapy.
Period: Overall Study
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy | Phase II: 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Phase II: Placebo Plus Standard IV Antibiotic Therapy
Started | 3 | 3 | 6 | 4 | 24 | 12
Completed | 2 | 3 | 5 | 4 | 21 | 12
Not Completed | 1 | 0 | 1 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 514G3 (2 mg/kg) Plus Standard IV Antibiotic Treatment: The participant received 514G3 (2 mg/kg) plus standard IV antibiotic treatment
- 514G3 (10 mg/kg) Plus Standard IV Antibiotic Treatment: The participant received 514G3 (10 mg/kg) plus standard IV antibiotic treatment
- 514G3 (40 mg/kg) Plus Standard IV Antibiotic Treatment: The participant received 514G3 (40 mg/kg) plus standard IV antibiotic treatment
- Placebo Plus Standard IV Antibiotic Treatment: The participant received placebo (sterile isotonic formulation buffered at pH 6.2 - 6.5) plus standard IV antibiotic treatment
- Phase II: 514G3 (40 mg/kg) Plus Standard IV Antibiotic Treatment: The participant received a single dose of 514G3 (40 mg/kg) plus standard IV antibiotic therapy
- Phase II: Placebo Plus Standard IV Antibiotic Treatment: The participant received a single dose of placebo plus standard IV antibiotic therapy.
- Total: Total of all reporting groups
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Treatment | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Treatment | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Treatment | Placebo Plus Standard IV Antibiotic Treatment | Phase II: 514G3 (40 mg/kg) Plus Standard IV Antibiotic Treatment | Phase II: Placebo Plus Standard IV Antibiotic Treatment | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 24 | 12 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 5 | 3 | 17 | 10 | 39
  >=65 years | 1 | 1 | 1 | 1 | 7 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 8 | 3 | 17
  Male | 1 | 2 | 4 | 3 | 16 | 9 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 5 | 2 | 13
  White | 2 | 2 | 4 | 2 | 14 | 9 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities
Description: Dose limiting Toxicity are defined as any Grade 3 or greater AE which is probably or definitely related to 514G3 occurring during the FU period after dosing. This measure determines and assesses the maximum tolerated dose (MTD) through participants who experienced DLT at different dose levels.
Time Frame: Pre-dose at Day 0 through Day 14. After day 14, samples are collected every other day including discharge, up to 30 days maximum
Population: Participants in Phase 1 who received a single IV dose of 514G3 (2mg/kg, 10mg/kg, and 40mg/kg) is a sequential manner
Measure: Number; unit: participants
Groups:
- 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received single dose of 2 mg/kg study drug (5143G) intravenously (IV) plus standard IV antibiotic therapy
- 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received single dose of 10 mg/kg study drug (5143G) intravenously (IV) plus standard IV antibiotic therapy.
- 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received single dose of 40 mg/kg study drug (5143G) intravenously (IV) plus standard IV antibiotic therapy.
- Placebo Plus Standard IV Antibiotic Therapy: A single dose of placebo plus IV antibiotic therapy
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy
Number analyzed (Participants) | 3 | 3 | 6 | 4
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced the Adverse Events
Description: A summary of SAEs and other non-serious AEs, regardless of causality
Time Frame: Adverse events occurring between day 0 and day 30 or hospital discharge whichever is shorter
Population: This measure assesses all adverse events from all randomized participants who received at least 1 dose of study drug according to the assigned treatment.
Measure: Number; unit: participants
Groups:
- Placebo Plus Standard IV Antibiotic Therapy: A single dose of placebo plus standard IV antibiotic therapy
- Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic Therapy: The participants received single dose of 40 mg/kg study drug (5143G) plus standard IV therapy
- Phase II: Placebo Plus Standard Intravenous Therapy: The participants received single dose of placebo with standard IV therapy
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic Therapy | Phase II: Placebo Plus Standard Intravenous Therapy
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 24 | 12
participants
  Serious adverse events | 1 | 1 | 1 | 2 | 5 | 5
  Non-serious adverse events | 2 | 3 | 6 | 4 | 23 | 9

3. Secondary Outcome: Time to Clearance of Bacteremia (Time to Sterile Culture From Date of Randomization)
Description: The time to sterile culture is the interval in days from the first dose of study drug until 2 consecutive days of negative blood cultures has occurred. The difference in this interval will be compared between patients randomized to placebo and those who received the highest dose of 514G3.
Time Frame: as for outcome 1
Population: All participants who had ≥1 positive blood cultures for staphylococcus Aureus within 2 days of randomization
Measure: Mean (Standard Deviation); unit: Days
Groups:
- 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received a single dose of 2 mg/kg study drug (5143G) intravenously (IV) plus standard IV antibiotic therapy.
- 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received a single dose of 10 mg/kg study drug (5143G) intravenously (IV) plus standard IV antibiotic therapy.
- 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy: The participants received a single dose of 40 mg/kg study drug (5143G) plus standard IV antibiotic therapy.
- Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic Treatment: The participants received single dose of 40 mg/kg study drug (5143G) plus standard IV therapy.
- Phase II: Placebo Plus Standard IV Antibiotic Therapy: The participants received single dose of placebo plus standard IV antibiotic therapy.
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic Treatment | Phase II: Placebo Plus Standard IV Antibiotic Therapy
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 24 | 12
Days | 1.67 (0.58) | 3.67 (1.53) | 2.0 (0.89) | 3.5 (1.91) | 2.54 (2.28) | 2.33 (1.50)

4. Secondary Outcome: Steady State Maximum Concentration of 514G3
Description: Blood samples were collected from participants who received study drug 514G3 for the determination of plasma concentration (Cmax).
Time Frame: as for outcome 1
Population: The PK-evaluable population included participants in the treatment arm who received 514G3 who had no major protocol violations and had documented adherence to the dosing and PK regimens. Data was not collected from subjects assigned to the placebo arm.
Measure: Mean (Standard Deviation); unit: microgram/millilitre
Groups:
- Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic: The participants received a single dose of 40 mg/kg study drug (5143G) plus standard IV therapy.
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic
Number analyzed (Participants) | 3 | 3 | 6 | 24
microgram/millilitre | 37.5 (22.4) | 198.0 (88.9) | 684.7 (143.1) | 740.0 (202.4)

5. Secondary Outcome: Length of Hospitalization (Duration of Hospitalization Stay After Randomization)
Description: This outcome measure assesses the impact of the treatment on the time that participants spend in the hospital. The duration of hospitalization is expressed as the average number of days hospitalized for all participants in their respective cohorts.
Time Frame: as for outcome 1
Population: The analysis population for this study will include all eligible subjects who have been randomized and received at least one dose of the study drug or placebo in both phases of the protocol.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Phase II: Placebo Plus Standard IV Antibiotic Therapy: The participants received a single dose of placebo plus standard IV antibiotic therapy.
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic | Phase II: Placebo Plus Standard IV Antibiotic Therapy
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 24 | 12
Days | 23.67 (21.36) | 11.33 (3.06) | 11.67 (4.18) | 20 (6.98) | 13.71 (9.07) | 17 (11.09)

6. Secondary Outcome: Difference in Opsonophagocytosis Activity Between Arms (Pharmacodynamics)
Description: Serum samples from patients will be assessed with an in-vitro Opsonophagocytosis assay which measures the ability of the serum to mediate uptake of staphylococcus aureus by white blood cells. Differences in the levels of activity will be compared between treatment and placebo. This outcome measure assesses the dose-dependent functional antibody response to 514G3, providing insights into its potential efficacy across different dosage levels compared to placebo. Higher titers in the drug-treated groups indicate better opsonophagocytic activity and thus better efficacy of the drug.
  Opsonophagocytosis activity (OPA) score quantifies the functional antibody response to the investigational drug 514G3.
  For Phase II, this score is determined using an Opsonophagocytosis assay and is calculated as follows:
  Relative Opsonophagocytosis activity = %Phagocytosis 30 minutes after treatment adjusted by baseline / %Phagocytosis of 500 ug/mL spike standard.
Time Frame: 14 days
Population: Safety population is all randomized participants who received at least one dose of the study treatment and provided valid Opsonophagocytosis assay (OPA) results'. Intent-to-treat (ITT) population is same as the safety population.
Measure: Mean (Standard Deviation); unit: percentage of phagocytosis activity
Arm/Group | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic | Phase II: Placebo Plus Standard IV Antibiotic Therapy
Number analyzed (Participants) | 24 | 12
percentage of phagocytosis activity | 129.7 (33.1) | 1.1 (2.5)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected between Day 0 and 30 days following the last administration of the investigational drug. This includes a follow-up period of 14 days after dosing to assess for Dose Limiting Toxicities (DLTs) and adverse events (AEs), with a Day 14 visit as an outpatient if the patient is discharged from the hospital prior to Day 14.
Groups:
- Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic: The participants received single dose of 40 mg/kg study drug (5143G) plus standard IV therapy.
Arm/Group | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy | Placebo Plus Standard IV Antibiotic Therapy | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic | Phase II: Placebo Plus Standard Intravenous Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/4 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/6 | 2/4 | 6/24 | 5/12
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 5/6 | 4/4 | 19/24 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy (N=3) | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy (N=3) | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy (N=6) | Placebo Plus Standard IV Antibiotic Therapy (N=4) | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic (N=24) | Phase II: Placebo Plus Standard Intravenous Therapy (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EMBOLIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — loss of perfusion to Left Lower Extremity resulting in Above Knee Amputation
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 514G3 (2 mg/kg) Plus Standard IV Antibiotic Therapy (N=3) | 514G3 (10 mg/kg) Plus Standard IV Antibiotic Therapy (N=3) | 514G3 (40 mg/kg) Plus Standard IV Antibiotic Therapy (N=6) | Placebo Plus Standard IV Antibiotic Therapy (N=4) | Phase II: 40 mg/kg Study Drug (514G3) Plus Standard IV Antibiotic (N=24) | Phase II: Placebo Plus Standard Intravenous Therapy (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute blood loss (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute on chronic congestive heart failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute post-operative respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 6 (12) | 2 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (6) | 3 (6) | 4 (5)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
BILATERAL AIRSPACE DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BILATERAL LEG OEDEMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SHOULDER PAIN BILATERAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD BILIRUBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION ACUTE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
PERINEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOMEGALY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COMMON COLD (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0)
BLOOD CALCIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GRIP STRENGTH DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DELIRIUM (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
COUGH DRY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (5) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
BLOOD NEUTROPHILS INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CHLORIDE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FIBRINOGEN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (12) | 2 (8)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
HYPERVOLAEMIA (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA HYPERVOLAEMIC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD ALBUMIN DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (14) | 1 (2)
BLOOD CALCIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (12) | 1 (3)
BLOOD CHLORIDE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 3 (4)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLOOD SODIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
BLOOD PHOSPHATE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD PROTEIN DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
THROMBOSIS VENA CAVA INFERIOR (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
BLOOD UREA DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
EPISTAXIS SEVERE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESSURE ULCER STAGE II (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
ALANINE AMINOTRANSFERASE DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD BICARBONATE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epidural abscess, paraspinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis injection site (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCLERAL ICTERUS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
POSTOPERATIVE RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Probable inflammatory myositis of serratus muscle, right
right arm and shoulder numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right Arm and Shoulder Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RIGHT CHEST WALL MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST WALL PAIN (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No